CLINICAL TRIAL: NCT05339399
Title: 4 Versus 6 cm Cervical os Dilatation to Demarcate Active Phase of Labour: Comparative Cross Ectional Study
Brief Title: 4 Versus 6 cm Active Phase of Labour
Status: Completed | Type: Observational
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Other Study IDs: FF-2021-173
Record Dates: First submitted 2022-04-06; First posted 2022-04-21 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Labor Complication; Cervix; Open
Keywords: active labour; 4 and 6 cm; low risk women
MeSH Terms: conditions — Obstetric Labor Complications; Uterine Cervical Incompetence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 4 cm cervical os dilatation: Low risk women with cervical os dilatation of 4 cm at amniotomy and whether they need oxytocin augmentation and analgesia.
  Interventions: Other: oxytocin augmentation
- 6 cm cervical os dilatation: Low risk women with cervical os dilatation of 6 cm at amniotomy and whether they need oxytocin augmentation and analgesia.
  Interventions: Other: oxytocin augmentation

INTERVENTIONS:
Other: oxytocin augmentation — Only observation of the outcome

SUMMARY:
A study to compare maternal and perinatal outcome between 4 and 6 cm cervical dilatation at amniotomy.

DETAILED DESCRIPTION:
Low risk women with singleton pregnancy are recruited. There are two groups which are 4 and 6 cm cervical os dilatation. The intrapartum management and labour outcomes are documented.

ELIGIBILITY:
Inclusion Criteria:

* singleton pregnancy
* no medical disorders
* no antenatal complications such as hypertension and diabetes

Exclusion Criteria:

* fetal anomaly
* one previous caesarean section
* other uterine scars

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Low risk pregnant women who delivers in our centre
Sampling Method: Non-Probability Sample
Enrollment: 155 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-02-10 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Caesarean section rate | from recruitment up to birth of neonate
  in percentage

SECONDARY OUTCOMES:
duration from amniotomy until delivery | from recruitment until up to delivery of neonate
  duration in minutes from recruitment until delivery
oxytocin augmentation | from recruitment until up to delivery of neonate
  percentage of those who required
Percentage of women with complications | from recruitment until up to 6 weeks post delivery
  complications such as postpartum haemorrhage and extended perineal tear
Percentage of neonates with complications | from birth of neonate up tom 7 days
  neonatal intensive care unit admission, Apgar score less than 7 at 5 minutes and cord pH <7.24

CONTACTS AND LOCATIONS:
Overall Officials: Rahana Abd Rahman, Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided